CLINICAL TRIAL: NCT04440774
Title: A Single Centre, Double-blind, Double-dummy Placebo-controlled, Randomised Phase Ib Study to Evaluate the Safety & Immunogenicity of the Candidate Chikungunya Vaccine ChAdOx1 Chik & the Zika Vaccine ChAdOx1 Zika in Healthy Adults in Mexico
Brief Title: Research Study to Assess New Chikungunya and Zika Vaccines in Healthy Adults in Mexico.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: CHIKA01
Record Dates: First submitted 2020-06-17; First posted 2020-06-22 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2021-09

CONDITIONS: Chikungunya; Zika
Keywords: Vaccine; ChAdOx1; Chikungunya; Zika; Mexico
MeSH Terms: conditions — Chikungunya Fever; Zika Virus Infection

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- CHIK low dose (Experimental): Volunteers will receive a single dose of 5x10^9 vp ChAdOx1 Chik delivered intramuscularly. Volunteers will be blinded and will not know if they have received the IMP or the placebo comparator
  Interventions: Biological: CHIK low dose
- CHIK mid dose (Experimental): Volunteers will receive a single dose of 2.5x10^10 vp ChAdOx1 Chik delivered intramuscularly. Volunteers will be blinded and will not know if they have received the IMP or the placebo comparator
  Interventions: Biological: CHIK mid dose
- CHIK high dose (Experimental): Volunteers will receive a single dose of 5x10^10 vp ChAdOx1 Chik delivered intramuscularly. Volunteers will be blinded and will not know if they have received the IMP or the placebo comparator
  Interventions: Biological: CHIK high dose
- ZIKA low dose (Experimental): Volunteers will receive a single dose of 5x10^9 vp ChAdOx1 Zika delivered intramuscularly. Volunteers will be blinded and will not know if they have received the IMP or the placebo comparator
  Interventions: Biological: ZIKA low dose
- ZIKA mid dose (Experimental): Volunteers will receive a single dose of 2.5x10^10 vp ChAdOx1 Zika delivered intramuscularly. Volunteers will be blinded and will not know if they have received the IMP or the placebo comparator
  Interventions: Biological: ZIKA mid dose
- ZIKA high dose (Experimental): Volunteers will receive a single dose of 5x10^10 vp ChAdOx1 Zika delivered intramuscularly. Volunteers will be blinded and will not know if they have received the IMP or the placebo comparator
  Interventions: Biological: ZIKA high dose
- CHIK ZIKA low dose (Experimental): Volunteers will receive a single dose of 5x10^9 vp ChAdOx1 Chik and 5x10^9 vp ChAdOx1 Zika delivered intramuscularly. Volunteers will be blinded and will not know if they have received the IMP or the placebo comparator
  Interventions: Biological: CHIK low dose; Biological: ZIKA low dose
- CHIK ZIKA mid dose (Experimental): Volunteers will receive a single dose of 2.5x10^10 vp ChAdOx1 Chik and 2.5x10^10 vp ChAdOx1 Zika delivered intramuscularly. Volunteers will be blinded and will not know if they have received the IMP or the placebo comparator
  Interventions: Biological: CHIK mid dose; Biological: ZIKA mid dose
- CHIK ZIKA high dose (Experimental): Volunteers will receive a single dose of 5x10^10 vp ChAdOx1 Chik and 5x10^10 vp ChAdOx1 Zika delivered intramuscularly. Volunteers will be blinded and will not know if they have received the IMP or the placebo comparator
  Interventions: Biological: CHIK high dose; Biological: ZIKA high dose
- Placebo (Placebo Comparator): Volunteers will receive a single dose of isotonic saline solution (0.9%) delivered intramuscularly. Volunteers will be blinded and will not know if they have received the IMP or the placebo comparator
  Interventions: Biological: Saline placebo

INTERVENTIONS:
Biological: CHIK low dose — A single dose of 5x10^9 vp ChAdOx1 Chik
  Arms: CHIK ZIKA low dose; CHIK low dose
Biological: CHIK mid dose — A single dose of 2.5x10^10 vp ChAdOx1 Chik
  Arms: CHIK ZIKA mid dose; CHIK mid dose
Biological: CHIK high dose — A single dose of 5x10^10 vp ChAdOx1 Chik
  Arms: CHIK ZIKA high dose; CHIK high dose
Biological: ZIKA low dose — A single dose of 5x10^9 vp ChAdOx1 Zika
  Arms: CHIK ZIKA low dose; ZIKA low dose
Biological: ZIKA mid dose — A single dose of 2.5x10^10 vp ChAdOx1 Zika
  Arms: CHIK ZIKA mid dose; ZIKA mid dose
Biological: ZIKA high dose — A single dose of 5x10^10 vp ChAdOx1 Zika
  Arms: CHIK ZIKA high dose; ZIKA high dose
Biological: Saline placebo — A single dose of isotonic saline solution (0.9%)
  Arms: Placebo

SUMMARY:
Phase Ib, single centre, double-blind, double-dummy placebo-controlled, randomised, stepwise dose escalated, vaccine trial to assess the safety and immunogenicity of the candidate ChAdOx1 Chik and ChAdOx1 Zika vaccines, given as a standalone vaccines or in co-administration. Healthy volunteers aged 18-50 years old, residents of the metropolitan area of Monterrey (Mexico), will be recruited as participants

DETAILED DESCRIPTION:
This trial consists of 4 intervention arms according to the vaccination product: 1) ChAdOx1 Chik, 2) ChAdOx1 Zika, 3) ChAdOx1 Chik and ChAdOx1 Zika as contralateral co-administration, and 4) placebo. There will be a total of 120 participants divided in ten study groups with 12 participants per group (Table 5.1). Groups 1 to 3 will receive ChAdOx1 Chik + placebo administered contralaterally, Groups 4 to 6 will receive ChAdOx1 Zika + placebo administered contralaterally, and Groups 7 to 9 will receive both ChAdOx1 Chik and ChAdOx1 Zika administered contralaterally. Group 10 will receive placebo in both arms.

Enrolment into this study will be implemented in a step-wise dose escalation manner. Participants will be first recruited into the vaccination groups at the lowest dose (Groups 1, 4 and 7). It is only after completion of these low dose groups and upon satisfactory interim clinical safety reviews that participants will be enrolled into the mid dose groups (Groups 2, 5 and 8). Participants in the high dose groups (Groups 3, 6 and 9) will be enrolled last, after completion and interim clinical safety reviews from the mid dose groups. Participants allocated to the Placebo group (Group 10) will be evenly distributed across the dose escalation model.

Randomisation procedures will be implemented accordingly, at a ratio of 3:3:3:1 for each of the four intervention arms.

The study involves a total of 9 visits (screening inclusive) and follow up will be undertaken for 6 months after vaccination day

Innovate UK (project number 971557)

ELIGIBILITY:
Inclusion Criteria:

1. Healthy men aged 18 to 50 (inclusive) years at the time of screening.
2. Healthy women aged 18 to 50 (inclusive) of child-bearing potential who agree to practice continuous effective contraception (see below) during the study and test negative for pregnancy on the day(s) of screening and vaccination.
3. Are residents of the metropolitan area of Monterrey, Nuevo León.
4. Provide written informed consent for participation in the study.
5. Able and willing (in the Investigator's opinion) to comply with all study requirements.
6. Agreement to inform study team of any impending vaccinations either before or during participation in the study.
7. Agreement to refrain from blood donation during the course of the study.
8. Agreement to refrain from receipt of any alphavirus or flavivirus vaccine throughout the duration of the study (e.g. investigational or licensed Yellow Fever, Japanese Encephalitis, Tick Borne Encephalitis or Dengue virus vaccines).

Exclusion Criteria:

1. Participation in another clinical trial in the 30 days preceding enrolment or during the study period.
2. Prior receipt of an investigational or licensed vaccine likely to impact on interpretation of the trial data (e.g. Adenovirus vectored vaccine, Chikungunya virus vaccine, Zika virus vaccine, Dengue virus vaccine).
3. Prior receipt of any vaccines administered ≤30 days before enrolment and/or planned during the during the study.
4. Administration of immunoglobulins and/or any blood products within the three months preceding the planned administration of the vaccine candidate.
5. Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (inhaled and topical steroids are allowed).
6. History of allergic disease or reactions likely to be exacerbated by any component of the vaccine. Any history of anaphylaxis in relation to vaccination.
7. History of autoimmune disease.
8. Any history of hereditary angioedema, acquired angioedema, or idiopathic angioedema.
9. Pregnancy, lactation or willingness/intention to become pregnant during the study.
10. History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ).
11. History of serious psychiatric condition likely to affect participation in the study
12. Bleeding disorder (eg. factor deficiency, coagulopathy or platelet disorder), or prior history of significant bleeding or bruising following IM injections or venepuncture.
13. Any other serious chronic illness requiring hospital specialist supervision at present or during the last 6 months.
14. Suspected or known current alcohol abuse. For men, intake greater than 5 drinks on a single occasion or more than 15 drinks per week; and for women, more than 4 drinks on a single occasion or more than 8 drinks per week. One drink =14 grams of pure alcohol.
15. Suspected or known injecting drug abuse in the 5 years preceding enrolment.
16. Seropositive for hepatitis B surface antigen (HBsAg).
17. Seropositive for hepatitis C virus (antibodies to HCV).
18. Any clinically significant abnormal finding on screening biochemistry or haematology blood tests or urinalysis.
19. Has history of chronic or acute severe neurologic condition. Including: Neurologic and Neuroinflammatory Disorders: ADEM, including site specific variants, Cranial Nerve Disorders (including paralyses/paresis), GBS (including Miller Fisher Syndrome and other variants), Immune-mediated Peripheral Neuropathies and Plexopathies, Optic Neuritis, Multiple Sclerosis, Narcolepsy, Transverse Myelitis, meningitis, or meningoencephalitis.
20. Any other significant disease, disorder or finding which may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data.
21. Seropositivity or cross-reactivity to Chikungunya virus, Zika virus or Dengue virus on screening tests.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2020-10-23 (Actual); Primary Completion 2022-02-18 (Actual); Study Completion 2022-02-18 (Actual)

PRIMARY OUTCOMES:
Assess the safety profile and tolerability of ChAdOx1 Chik and ChAdOx1 Zika in healthy participants: occurrence of local reactogenicity signs and symptoms | 7 days post vaccination
  Occurrence of solicited local reactogenicity signs and symptoms for 7 days following vaccination.
Assess the safety profile and tolerability of ChAdOx1 Chik and ChAdOx1 Zika in healthy participants: occurrence of solicited systemic reactogenicity signs and symptoms | 7 days post vaccination
  Occurrence of solicited systemic reactogenicity signs and symptoms for 7 days following the vaccination.
Assess the safety profile and tolerability of ChAdOx1 Chik and ChAdOx1 Zika in healthy participants: occurrence of unsolicited adverse events | 28 days post vaccination
  Occurrence of unsolicited adverse events for 28 days following vaccination
Assess the safety profile and tolerability of ChAdOx1 Chik and ChAdOx1 Zika in healthy participants through standard blood tests (full blood count, liver and kidney function tests) | 28 days post vaccination
  Change from baseline for safety laboratory measures (haematology and biochemistry blood results)
Assess the safety profile and tolerability of ChAdOx1 Chik and ChAdOx1 Zika in healthy participants: occurrence of serious adverse events during the whole study duration | 6 months post vaccination
  Occurrence of serious adverse events during the whole study duration

SECONDARY OUTCOMES:
Assess the humoral immunogenicity of the candidate vaccines ChAdOx1 Chik and ChAdOx1 Zika via PRNT50 | 6 months post vaccination
  Plaque-reduction neutralisation tests at 50% (PRNT50) against chikungunya and Zika virus.
Assess the humoral immunogenicity of the candidate vaccines ChAdOx1 Chik and ChAdOx1 Zika via IgG ELISA antibody titres | 6 months post vaccination
  IgG ELISA antibody titres against proteins of Chikungunya and Zika virus

CONTACTS AND LOCATIONS:
Overall Officials: Abiel Homero Mascareñas de los Santos, MD, Principal Investigator — Hospital Universitario "Dr. José Eleuterio González" Universidad Autónoma de Nuevo León
Locations (1):
- Hospital Universitario "Dr. José Eleuterio González" de la Universidad Autónoma de Nuevo León., Monterrey, Nuevo León, Mexico